CLINICAL TRIAL: NCT03327077
Title: Music in Urgent and Emergent Settings (MUES) Trial: Phase Three
Brief Title: Music in Urgent and Emergent Settings
Acronym: MUES III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Endowment for the Arts, United States (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB201700938; 15-3800-7018 (Other Grant/Funding Number: US National Endowment for the Arts)
Record Dates: First submitted 2017-10-26; First posted 2017-10-31 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Musculoskeletal Pain
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention)
- Intervention Group (Experimental): Music group
  Interventions: Other: Live Preferential Music

INTERVENTIONS:
Other: Live Preferential Music — Trained musicians will play live preferential music to ED patients who consent to participate.
  Arms: Intervention Group

SUMMARY:
The purpose of this study is to study the impact of Live Preferential Music on the patient perception of pain and management of pain syndromes in the ED.

DETAILED DESCRIPTION:
The purpose of this study is to study the impact of Live Preferential Music on the patient perception of pain and management of pain syndromes in the ED. This study follows a prospective experimental design where patients will be assigned to two groups: one that receives the music intervention and one that does not receive music intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥18
2. Chief complaint of musculoskeletal pain
3. Gender: Male or Female
4. Ethnicity: Any
5. Physical ability: Any
6. Language: English
7. Cognitive skill/education: grade 2 reading level or above
8. Physically and cognitively able to participate in study procedures

Exclusion Criteria:

1. Patients who are unable to participate in the informed consent process
2. Prisoners

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Pain reduction | 60 to 90 minutes

SECONDARY OUTCOMES:
Cost of care | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Tyndall, MD, Principal Investigator — University of Florida
Locations (1):
- Unversity of Florida, Gainesville, Florida, United States